CLINICAL TRIAL: NCT04479969
Title: Enabling Independent Living by Expanding Access to Home-Based Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-003806; 1R43HL151461 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): This is a small study to assess the usability of video conferencing. A total of 10 patients will be enrolled, 5 of which will be Spanish speakers. All patients will test the video conferencing.
  Interventions: Behavioral: Video Chat

INTERVENTIONS:
Behavioral: Video Chat — Video chat with health coach using a computer tablet.

SUMMARY:
The purpose of this study is to test an existing home-based pulmonary rehab program with the addition of video chat and a capability of a Spanish version.

DETAILED DESCRIPTION:
The purpose of this research is to test video chat on a computer tablet that is used for Pulmonary Rehabilitation. We are interested in learning patients' thoughts on how easy or difficult video chat is to use and the translation to Spanish and the feed back from Spanish speaking patients .

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 40 years old.
* Patients mist have a diagnosis of GOLD stage II, III, or IV COPD documented by pulmonary function testing.
* Patients must be a current or previous smoker with at least 10 pack-years of cigarette smoking.

Additional Inclusion Criteria to test Spanish version of system:

* Be a native Spanish speaker.

Exclusion Criteria:

* Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency).
* Patients planning to move out of the state or who are not living in the healthcare area.
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Qualitative Interview | Week 1
  A Qualitative Interview will be conducted over the phone asking about the video chat experience.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials